CLINICAL TRIAL: NCT02270801
Title: Recombinant Human Thrombopoietin (rhTPO) in Management of Immune Thrombocytopenia (ITP)in Pregnancy: a Single-center Clinical Trial
Brief Title: Recombinant Human Thrombopoietin (rhTPO) in Management of Immune Thrombocytopenia (ITP) in Pregnancy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rhTPO-ITP-Pregnancy
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-03

CONDITIONS: Immune Thrombocytopenia; Pregnancy
Keywords: recombinant human thrombopoietin; immune thrombocytopenia; pregnancy
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rhTPO (Experimental): rhTPO will be given intravenously at a dose of 300U/kg every day. Dose will be tapered to 300U/kg every other day when platelet count rise over 50×10^9/L. Maintenance will be continued after delivery and the dose will be further reduced to 300U/kg per week.
  Interventions: Drug: rhTPO

INTERVENTIONS:
Drug: rhTPO — rhTPO will be given intravenously at a dose of 300U/kg every day. Dose will be tapered to 300U/kg every other day when platelet count rise over 50×10^9/L. Maintenance will be continued after delivery and the dose will be further reduced to 300U/kg per week.
  Other Names: TPIAO; S20050048/49 (SFDA, China)

SUMMARY:
This clinical trial is undertaking by Qilu Hospital of Shandong University, aims at evaluating efficacy and safety of rhTPO in management of ITP in pregnancy.

DETAILED DESCRIPTION:
The investigators are undertaking a single-center, non-randomized, non-controlled trial of 30 ITP patients in pregnancy from Qilu Hospital of Shandong University. ITP patients in pregnancy who failed to respond to prednisone, IVIG and developed refractoriness to platelet transfusion will be given rhTPO intravenously at a dose of 300U/kg every day. Dose will be tapered to 300U/kg every other day when platelet count rise over 50×10^9/L. Maintenance will be continued after delivery and the dose will be further reduced to 300U/kg per week. Platelet count, bleeding and other symptoms will be evaluated before and after treatment. Adverse events will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18-50 years old.
2. After 12 weeks gestation.
3. Diagnosed with ITP meeting the diagnostic criteria for immune thrombocytopenia.
4. Patients who have no response or relapsed after Corticosteroid or IVIG.
5. Patients developed refractoriness to platelet transfusion.
6. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
7. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit.
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
4. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
5. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
6. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Early Response | one month after delivery
  Response rate (CR+R) at the 14th day, the 10th week from the initial injection of rhTPO, ante partum and one month after delivery. CR is defined as platelet count ≥ 100×109/L, and R is defined as platelet count of >30×109/L with at least a doubling of the baseline value.

SECONDARY OUTCOMES:
Safety | six months after delivery
  Adverse events in patients and infants.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD PhD, Principal Investigator — Shandong University
Locations (1):
- Shandong University Qilu hospital, Jinan, Shandong, China